CLINICAL TRIAL: NCT02877888
Title: A Randomised Controlled Trial to Measure Effectiveness of Sodium Fluoride Varnish to Prevent Dental Caries in School Children Between Age of 6 and 7 Years
Brief Title: Effectiveness of Fluoride Varnish in Prevention of Dental Caries in School Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Peradeniya (Other)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Dr. RM Jayasinghe, senior lecturer, University of Peradeniya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FRC/FDS/UOP-2014/25
Record Dates: First submitted 2016-08-11; First posted 2016-08-24 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Dental Caries
Keywords: cost effectiveness; fluoride varnish; dental caries
MeSH Terms: conditions — Dental Caries | interventions — sodium fluoride topical preparation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- drug fluoride varnish /strength 22600ppm (Experimental): intervention: drug :fluoride varnish 22600ppm topical application every 6 months for a total period of 2 years
  Interventions: Drug: fluoride varnish 22600ppm
- placebo comparator (No Intervention): placebo:use of routine dental advice

INTERVENTIONS:
Drug: fluoride varnish 22600ppm — topical application on teeth every 6months
  Other Names: 5% duraphat
  Arms: drug fluoride varnish /strength 22600ppm

SUMMARY:
Despite the availability of free health dental service in Sri Lanka, the prevalence and severity of dental caries among 6year old school children stand at a very high level according to the results of national oral health survey in 1983/84, 94/95 and 2002/2003. Professional fluoride varnish application has become popular as variety of studies has found that it is an efficient method in reducing dental caries. The simplicity of its application makes it very suitable and practical for use in dental clinics and outreach dental services, especially in young children.

Aim of this study is to evaluate the cost effectiveness of 6 monthly application of sodium fluoride varnish in prevention of dental caries in permanent incisors and molars in children between 6 and 7 years in a suburban setting in Sri Lanka. This will be a double-blind, randomized controlled trial. A sample of school children (6-7 years) will be randomized into varnish and control groups. All the children will receive routine caries preventive measures of oral hygiene instructions, dietary advice and professional cleaning. Children in varnish group will receive fluoride varnish professionally applied after prophylaxis every 6 months. Clinical examinations of all children will be performed at the beginning of the study and 1 year and 2 years later. All the caries at the dentinal level of both groups will be stabilized with temporary restorations at the beginning. During this period, each school will be visited four times at 6-month interval for recruitment, dental examinations, and fluoride varnish applications. Recruited children will be randomly assigned to either a treatment (5% NaF varnish) or a control group. Caries examinations will be conducted using the International Caries Detection and Assessment System (ICDAS). The cost for the dental team's school visits; cost involved in the treatment of dental caries throughout the course of the study in both groups will be evaluated and compared at the end of the study. The sample size is calculated as 160 each arm to detect 5% caries change with 80% power. Analysis The effect of intervention will be measured by number of caries prevented. New caries in the usual care and intervention group will be calculated after the completion of the study. The costs for intervention will be estimated. The costs will be estimated for the dental material, time for human resources and indirect costs.

DETAILED DESCRIPTION:
Background

Dental caries remains a significant public health problem with socioeconomic, dietary and microbiological factors playing a major role as risk factors in initiation and progression of the disease. It is the most common cause of toothache and hospital admissions in young children. Dental caries in school children not only causes pain, but also impacts school attendance, parents' work hours, children's ability to eat, play and sleep. Therefore, dental caries when present significantly reduces the health related quality of life of a child.

Evidence-based studies indicate oral health prevention is cost-effective and saves children from pain and lost days of school.Therefore the measures taken to prevent the develop¬ment of dental caries could include bacterial biofilm control, dietary counselling, fluoride toothpastes, mouth rinses, varnishes, gels and foams, and casein-derived remineralisation pastes and placing resin-based/glass-ionomer pit and fissure sealants. ) Professional fluoride varnish application has become popular as variety of studies has discussed its effect in reducing dental caries.

Fluoride varnish was incorporated into clinical dentistry to reduce caries; its use in the U.S. has increased progressively since it was approved by the FDA in 1994. Fluoride varnish's effectiveness in caries prevention, ease of application, and safety give it an advantage over other types of topical fluoride treatments (such as gels and rinses) or other caries management methods. As a result, it is regarded as one of the superior topical fluoride agents for young children. Fluoride varnish also prolongs the contact time between fluoride and tooth surface to reduce caries. Its active ingredient is usually 5% sodium fluoride, or 22,600 ppm fluoride. It also has recently gained much attention in dentistry because the risk of dental fluorosis is also minimal.The simplicity of its application makes it very suitable and practical for use in dental clinics and outreach dental services, especially in young children and in other special needs groups.

Justification

Despite the availability of free health dental service in Sri Lanka, the prevalence and severity of dental caries among six and seven years old school children in Sri Lanka stand at a very high level according to the results of national oral health survey in 1983/84, 94/95 and 2002/2003. The prevalence is 78% (83/84), 76.4% (94/95) and 65.5% (2002/2003) whereas the dmft is 4.4, 4.1 and 3.6.

The simplicity of its application makes it very suitable and practical for use in dental clinics and outreach dental services, especially in young children and in other special needs groups.

Up to date there is no other study carried out on cost effectiveness of fluoride varnish application on teeth in Sri Lankan population. Therefore, the results of the study will be beneficial in implementation and identification of advantages of fluoride varnish application on teeth in young children.

Aim

the main objective of this study was to evaluate the effectiveness of six monthly application of sodium fluoride varnish in prevention of dental caries in deciduous teeth, permanent incisors and molars in children between six and seven years in Sri Lanka.

The specific objective is:

1. To find out the association between dental caries and the social status of the child (e.g. mother's education, father's education, monthly family income etc.)

Methods

This was a double-blind, randomized controlled trial. The study has been registered with clinical trials registry (NCT02877888).

The study population was school children aged six to seven years, living in Kurunegala district. The inclusion and exclusion criteria used in the study are described below. The study was conducted at Maliyadeva Adarsha Vidyalaya and Wayamba Royal college, Kurunegala from month year to month year. The sample was selected according to below criteria…

Inclusion Criteria:

* Children with at least one permanent tooth present.
* Age 6 to 7 years. Children under 6 years of age were enrolled in the study if at least one permanent tooth has erupted.
* Residing in Kurunegala municipal council region and tap water is consumed (fluoride levels in drinking water was considered similar).

Exclusion Criteria:

* Children with ulcerative gingivitis and stomatitis. (These children were referred for treatment.)
* No permanent tooth present or stainless steel crowns only.

The students meeting the inclusion and exclusion criteria was randomly assigned, using block randomization in blocks of four, using a computer generated set of random numbers, to either varnish (5% Sodium Fluoride) or control group. A set of random numbers was used to create an allocation sequence, which was contained in individual opaque envelopes for used by the chief investigator. As the patients were recruited, the next envelope in the sequence was opened and the student was assigned to the stated group. All randomisation, sequence generation, and preparation of group allocation materials was performed by a third party who had no direct contact with the clinical aspects of the trial.

The sample size was calculated as 160 each arm to detect 5% caries change with 80% power. All children in both groups were provided with a self-administered pre tested questionnaire to assess the quality of life associated with presence of dental caries. Further, all the children received routine caries preventive measures of oral hygiene instructions, dietary advice and professional cleaning. Clinical examinations of all children were performed at the beginning of the study and 1 year and 2 years later. All the caries at the dentinal level of both groups were stabilized with temporary restorations at the beginning. Both varnish and control groups were subjected to use of fluoride tooth paste of 1000ppm. Children in the intervention group received fluoride varnish professionally applied after prophylaxis every 6 months combined with counselling on maintenance of oral hygiene and diet for a period of 2 years. The control group was only subjected to counselling on maintenance of oral hygiene and diet.

During the period of two years, a team visited each school four times at six months' interval for recruitment, dental examinations, and fluoride varnish applications. Trained interviewers collected data on oral health habits and sociodemographic characteristics of the children. Caries examinations were conducted using the International Caries Detection and Assessment System (ICDAS).

The primary outcome studied was the number of new caries in the two study groups. Students and the interviewers were blinded to the intervention (varnish application or control) and they were blinded to the hypothesis, which was investigated in this study.

Analysis

The mean number of caries between different groups, segregated according to the variables assessed in the study, were compared. The mean number of caries in a particular group was calculated by dividing the total number of caries in a particular group by the total number of students in that group. As the number of caries showed a skewed distribution, Mann-Whitney U test was used compare the groups. Level of significance was considered as p<0.05.

The effect of intervention was measured by the mean number of new caries in different groups. The number of new caries in the usual care and intervention group was calculated at each time point of the survey. The mean number of new caries between the two groups were compared using Mann-Whitney U test. To assess the independent effect of the intervention on the incidence of caries, when other factors are controlled, multiple linear regression was applied.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least one permanent tooth present.
* Age 6 to 7 years. Children under 6 years of age may be enrolled in the study if at least one permanent tooth has erupted.
* Residing in Kurunegala municipal council region and tap water is consumed (fluoride levels in drinking water is normal).
* Parental consent must be provided. If the parent is not the primary caregiver, a legal guardian or a family member who is the primary care provider must sign the consent form.

Exclusion Criteria:

* Children with ulcerative gingivitis and stomatitis. (These children will be referred for treatment.)
* No permanent teeth present or stainless steel crowns only.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
number of caries prevented in the intervention and control gropus | every 6 months for 2 years
  Association between sodium fluoride varnish application and the mean number of new dental caries atdifferent points are shown in table 3.
  Table 3: Association between sodium fluoride varnish application and new dental caries at different time points
  Period Mean number of dental caries in the Intervention Group Mean number of dental caries in the Control Group p value# 2015 May 0.94 1.79 <0.001 2015 Dec 1.69 1.77 <0.001 2016 Nov 1.50 1.97 <0.001
  #Mann-Whitney U test
Relationship of quality of life of children with dental caries and without dental caries | at the beginning of study after examination
  The total sample consisted of 321 students, with 161 and 162 in control and intervention groups respectively. Mean number of caries was significantly high among those who had difficulty in chewing, difficulty in vigorous chewing, difficulty in taking hot or cold food.
  Percentage of students with at least one dental caries at the beginning of the study was compared between different variables. If a student had at least one tooth with dental caries, was taken as positive for dental caries. Of the total population 115 (65.7%) of the students in the 6 age group had at least one tooth with dental caries and equal proportion was found among those who were more than six years as well. Difficulty in chewing (<0.001), difficulty chewing vigorously (<0.001), difficulty taking cold or hot food (<0.001) and difficulty taking sweets (0.034) were experienced more by the students who had at least one dental caries.

SECONDARY OUTCOMES:
Independent association between vanish intervention and new dental caries | every 6 months for 2 years
  To assess the independent effect of the intervention on development of new dental caries, when other factors are controlled, multiple linear regression was applied. Application of vanish was significantly associated with less number of new dental caries at two time points (May 2015 and Nov 2016) of the survey.
  Period β coefficient 95% CI p value May 2015 Intervention -0.84 -1.24 - -0.45 <0.001 Control 1 Dec 2015 Intervention 0.09 -0.45 - 0.64 0.733 Control 1 Nov 2016 Intervention -0.49 -1.0 - -0.28 0.043 Control 1

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Academy on Pediatric Dentistry; American Academy of Pediatrics. Policy on early childhood caries (ECC): classifications, consequences, and preventive strategies. Pediatr Dent. 2008-2009;30(7 Suppl):40-3. No abstract available. PMID 19216381
- [Background] Gugwad SC, Shah P, Lodaya R, Bhat C, Tandon P, Choudhari S, Patil S. Caries prevention effect of intensive application of sodium fluoride varnish in molars in children between age 6 and 7 years. J Contemp Dent Pract. 2011 Nov 1;12(6):408-13. doi: 10.5005/jp-journals-10024-1068. PMID 22269229
- [Background] Liu BY, Lo EC, Chu CH, Lin HC. Randomized trial on fluorides and sealants for fissure caries prevention. J Dent Res. 2012 Aug;91(8):753-8. doi: 10.1177/0022034512452278. Epub 2012 Jun 26. PMID 22736448
- [Background] Chu CH, Lo E. Uses of sodium fluoride varnish in dental practice. Ann R Australas Coll Dent Surg. 2008 Jun;19:58-61. PMID 19728633
- [Background] Tickle M, Milsom KM, Donaldson M, Killough S, O'Neill C, Crealey G, Sutton M, Noble S, Greer M, Worthington HV. Protocol for Northern Ireland Caries Prevention in Practice Trial (NIC-PIP) trial: a randomised controlled trial to measure the effects and costs of a dental caries prevention regime for young children attending primary care dental services. BMC Oral Health. 2011 Oct 10;11:27. doi: 10.1186/1472-6831-11-27. PMID 21985746
- [Background] Lewis CW, Johnston BD, Linsenmeyar KA, Williams A, Mouradian W. Preventive dental care for children in the United States: a national perspective. Pediatrics. 2007 Mar;119(3):e544-53. doi: 10.1542/peds.2006-1958. PMID 17332174
- [Background] Greig V, Conway DI. Fluoride varnish was effective at reducing caries on high caries risk school children in rural Brazil. Evid Based Dent. 2012;13(3):78-9. doi: 10.1038/sj.ebd.6400874. PMID 23059920
- [Background] Bali RK, Mathur VB, Talwar PP, Chanana HB. National Oral Health Survey and Fluoride Mapping, 2002-2003, India. Delhi: Dental Council of India; 2004
- [Background] Child Dental Health Survey 2013: England, Wales and Nothern Ireland 2013
- [Background] State Oral Health Surveys. Centers for Disease Control and Prevention 2018
- [Result] Chu CH, Lo EC. A review of sodium fluoride varnish. Gen Dent. 2006 Jul-Aug;54(4):247-53. PMID 16903196
- [Result] Dimitropoulos Y, Holden A, Gwynne K, Irving M, Binge N, Blinkhorn A. An assessment of strategies to control dental caries in Aboriginal children living in rural and remote communities in New South Wales, Australia. BMC Oral Health. 2018 Oct 29;18(1):177. doi: 10.1186/s12903-018-0643-y. PMID 30373592
- [Result] James P, Parnell C, Whelton H. The caries-preventive effect of chlorhexidine varnish in children and adolescents: a systematic review. Caries Res. 2010;44(4):333-40. doi: 10.1159/000315346. Epub 2010 Jul 7. PMID 20606432
- [Result] Moberg Skold U, Petersson LG, Lith A, Birkhed D. Effect of school-based fluoride varnish programmes on approximal caries in adolescents from different caries risk areas. Caries Res. 2005 Jul-Aug;39(4):273-9. doi: 10.1159/000084833. PMID 15942186
- [Result] Neidell M, Shearer B, Lamster IB. Cost-Effectiveness Analysis of Dental Sealants versus Fluoride Varnish in a School-Based Setting. Caries Res. 2016;50 Suppl 1:78-82. doi: 10.1159/000439091. Epub 2016 Apr 22. PMID 27100884